CLINICAL TRIAL: NCT00342810
Title: Continued Analyses of Epidemiologic Risk Factors Using Existing Framingham Eye and Heart Study Data
Brief Title: Analyses of Existing Framingham Data
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903232; 03-EI-N232
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-04-25

CONDITIONS: Eye Diseases
Keywords: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Since 1948, the Framingham Study has examined a group of men and women every two years for the primary purpose of studying the incidence and prevalence of cardiovascular disease and its risk factors. In 1971 the Framingham Study began a study of the offspring of the original group, including data collection on blood pressure, cigarette smoking, weight, and other factors that are of interest to studies of eye disease. Researchers gave eye exams to some of the original group and to the offspring group. Data from these eye exams have been used to examine risk factors for cataracts, diabetic retinopathy, myopia, and glaucoma.

The purpose of this study is to use the previously collected data for continued research on eye-related disorders. No new eye examinations will be conducted.

...

DETAILED DESCRIPTION:
We propose to continue to analyze existing Framingham Eye and Heart Study data to identify possible risk factors for various eye diseases. Originally begun in 1948 by the National Heart, Lung and Blood Institute (NHLBI), the Framingham Heart Study has been examining a population-based cohort of men and women biennially since 1948 for the primary purpose of studying the incidence and prevalence of cardiovascular disease and its risk factors. In 1971 the Heart Study began a prospective study of the offspring of the original cohort. The Heart Study has collected data on blood pressure, cigarette smoking, weight and many other factors of interest for epidemiologic studies of eye disease. Eye examinations were conducted on the survivors of the original cohort in a collaborative effort between the NEI and the NHLBI between 1973 and 1975 (Framingham Eye Study I; FES I) and then again between 1986 and 1989 (Framingham Eye Study II; FES II). Eye examinations were conducted on the Offspring Cohort from 1989 to 1991 (Framingham Offspring Eye Study; FOES). The Framingham data are unique in allowing epidemiologic studies with both cross sectional and longitudinal designs. Over the years, data from the Heart Study and the various eye studies have been used to examine demographic and risk factor characteristics for cataract, diabetic retinopathy, myopia, and glaucoma. To date this collaborative effort has yielded 31 publications by the National Eye Institute's Division of Epidemiology and Clinical Research; Rita Hiller is an author of 11. This proposal is for the continued use of the previously collected Framingham data. All studies will be done in collaboration with Heart Study investigators from Boston University which manages the study and conducts annual IRB reviews. No new eye examinations will be done.

ELIGIBILITY:
* This study is of existing ocular data from the Framingham Eye Study. Since the participants have already been recruited, there are no further exclusions from the study.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6061 (Actual)
Dates: Start 2003-06-25; Study Completion 2018-04-25

PRIMARY OUTCOMES:
Explore associations using study data | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vitale, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Eye Institute (NEI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ederer F, Hiller R, Taylor HR. Senile lens changes and diabetes in two population studies. Am J Ophthalmol. 1981 Mar;91(3):381-95. doi: 10.1016/0002-9394(81)90293-2. PMID 7211996
- [Background] Sperduto RD, Hiller R. The prevalence of nuclear, cortical, and posterior subcapsular lens opacities in a general population sample. Ophthalmology. 1984 Jul;91(7):815-8. doi: 10.1016/s0161-6420(84)34233-6. PMID 6472815
- [Background] Hiller R, Sperduto RD, Podgor MJ, Ferris FL 3rd, Wilson PW. Diabetic retinopathy and cardiovascular disease in type II diabetics. The Framingham Heart Study and the Framingham Eye Study. Am J Epidemiol. 1988 Aug;128(2):402-9. doi: 10.1093/oxfordjournals.aje.a114980. PMID 3293436